CLINICAL TRIAL: NCT05513872
Title: A Mechanistic Test of Treatment Strategies to Foster Practice Quitting
Brief Title: Overcoming Nicotine Dependence to Enable Quitting
Acronym: ON-DEQ
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Rush University Medical Center (Other)
Collaborators: Medical University of South Carolina (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 20121702
Record Dates: First submitted 2022-08-16; First posted 2022-08-24 (Actual); Last update posted 2025-08-17 (Actual); Status verified 2025-08

CONDITIONS: Tobacco Use; Smoking Cessation; Smoking Behaviors; Nicotine Dependence; Nicotine Withdrawal
Keywords: tobacco; smoking cessation; nicotine dependence; nicotine replacement therapy; behavioral treatment
MeSH Terms: conditions — Tobacco Use; Smoking Cessation; Smoking; Tobacco Use Disorder | interventions — Nicotine Replacement Therapy; Counseling; Motivational Interviewing

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- Condition #1 (Experimental): NRT Sampling = On Behavioral Counseling = Practice Quitting
  Interventions: Drug: Nicotine Replacement Therapy (NRT) Sampling; Behavioral: Practice Quitting (PQ) Counseling
- Condition #2 (Experimental): NRT Sampling = Off Behavioral Counseling = Practice Quitting
  Interventions: Behavioral: Practice Quitting (PQ) Counseling
- Condition #3 (Experimental): NRT sampling = On Behavioral counseling = Motivational Interviewing
  Interventions: Drug: Nicotine Replacement Therapy (NRT) Sampling; Behavioral: Motivational Interviewing (MI) Counseling
- Condition #4 (Experimental): NRT sampling = Off Behavioral counseling = Motivational Interviewing
  Interventions: Behavioral: Motivational Interviewing (MI) Counseling

INTERVENTIONS:
Drug: Nicotine Replacement Therapy (NRT) Sampling — Participants randomized to this condition will receive a 4-week nicotine replacement therapy (NRT) starter kit containing both nicotine lozenges and patches in their original packaging.
  Arms: Condition #1; Condition #3
Behavioral: Practice Quitting (PQ) Counseling — Practice Quitting (PQ) counseling will consist of four weekly treatment sessions, with an initial 45-minute session followed by three 20-minute sessions. The goals of the counseling sessions are 1) to gradually expose patients to nicotine withdrawal symptoms through practice quitting, and 2) to reduce fear and avoidance of the physical sensations associated with nicotine withdrawal.
  Arms: Condition #1; Condition #2
Behavioral: Motivational Interviewing (MI) Counseling — Motivational Interviewing (MI) counseling will consist of four weekly treatment sessions, with an initial 45-minute session followed by three 20-minute sessions. Counseling content will incorporate MI-consistent principles, such as open questions, simple and complex reflections, and affirmations to facilitate participant statements in favor of behavior change. Discussion will focus on the motivational topics outlined in the USPHS guidelines for smokers not ready to quit: 1) relevance of smoking cessation or reduction to the individual, 2) risks of continued heavy smoking, 3) rewards of quitting and reduction, and 4) roadblocks to success, on a 5) repeated basis.
  Arms: Condition #3; Condition #4

SUMMARY:
Tobacco use disorder is a chronic, relapsing health condition that necessitates a chronic care approach. However, traditional smoking cessation treatment programs allocate nearly all their resources only to those smokers who are willing to set a quit date. This is problematic because few smokers are ready to set a quit date at any given time, and a smoker's stated intention to quit can change rapidly.

One novel potential treatment strategy is to foster practice quitting (PQ), defined as attempting to not smoke for a few hours or days, without pressure or expectation to permanently quit. Although a growing body of evidence supports the role of practice quitting in fostering permanent quit attempts and cessation, there is a significant knowledge gap regarding which treatment strategies should be used to engage smokers in practice quitting. The proposed study will test the role of PQ counseling vs. Motivational Interviewing (MI) counseling, and NRT sampling (four-week supply of nicotine lozenges and patches) vs. none.

DETAILED DESCRIPTION:
Tobacco use disorder is a chronic, relapsing health condition that necessitates a chronic care approach. However, traditional smoking cessation treatment programs allocate nearly all their resources only to those smokers who are willing to set a quit date. This is problematic because few smokers are ready to set a quit date at any given time, and a smoker's stated intention to quit can change rapidly.

One novel potential treatment strategy is to foster practice quitting (PQ), defined as attempting to not smoke for a few hours or days, without pressure or expectation to permanently quit. Practice quitting represents a useful treatment exercise, as it offers a point of focus for behavior change coaching and goal-setting, with or without a planned quit date. The proposed study will test the role of PQ counseling vs. Motivational Interviewing (MI) counseling, and NRT sampling (four-week supply of nicotine lozenges and patches) vs. none. Specific aims are to:

Aim 1: Evaluate hypothesized mechanisms of action for PQ counseling and NRT sampling on incidence of quit attempts by 6 months among current smokers who are not planning to quit in the next 30 days (N=780). We will test the mediational effect of each variable on the relationship between PQ-focused treatment and incidence of quit attempts.

Aim 2: Test both the individual and combined roles of PQ counseling and NRT sampling on incidence of quit attempts by 6 months. We hypothesize that PQ counseling combined with NRT sampling will produce the highest rates of quit attempts through an additive relationship between these two treatment components.

ELIGIBILITY:
Inclusion Criteria:

Eligible participants will be males and females who:

1. are 18 years or older
2. report current daily cigarette smoking (≥ 5 cigarettes per day)
3. are not planning to quit in the next 30 days
4. are not currently engaged in smoking cessation treatment
5. are motivated to quit or engage in a non-cessation goal (i.e., reduce smoking, learn more about treatment options, and/ or try out skills to change smoking) in the next 6 months
6. are English speaking
7. reside in the continental United States
8. have access to a smartphone that can be used to complete study procedures

Exclusion Criteria:

Participants will be excluded for daily vaping/ electronic cigarettes use (i.e., use for ≥ 25 days within past 30 days) and any FDA contraindications for NRT use if they:

1. are pregnant/breastfeeding
2. had recent cardiovascular trauma such as myocardial infarction
3. had a stroke within the past 3 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 780 (Estimated)
Dates: Start 2023-03-24 (Actual); Primary Completion 2027-08-30 (Estimated); Study Completion 2027-08-30 (Estimated)

PRIMARY OUTCOMES:
Any incidence of a quit attempt | At 6-month follow-up assessment
  Intentional abstinence of ≥ 24 hours between the end of treatment and the 6-month follow-up assessment

SECONDARY OUTCOMES:
Abstinence status at 1-month follow-up | At 1-month follow-up assessment
  Self-report of no smoking (not even a puff) within the previous 7 days, confirmed by an expired carbon monoxide (CO) reading of ≤ 6 parts per million (ppm).
Abstinence status at 3-month follow-up | At 3-month follow-up assessment
  Self-report of no smoking (not even a puff) within the previous 7 days, confirmed by an expired carbon monoxide (CO) reading of ≤ 6 parts per million (ppm).
Abstinence status at 6-month follow-up | At 6-month follow-up assessment
  Self-report of no smoking (not even a puff) within the previous 7 days, confirmed by an expired carbon monoxide (CO) reading of ≤ 6 parts per million (ppm).

CONTACTS AND LOCATIONS:
Overall Officials: Amanda Mathew, PhD, Principal Investigator — Rush University Medical Center
Locations (1):
- Rush University Medical Center, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No